CLINICAL TRIAL: NCT04483960
Title: A Multi-centre Randomised Adaptive Platform Clinical Trial to Assess Clinical, Virological and Immunological Outcomes in Patients With SARS-CoV-2 Infection (COVID-19)
Brief Title: Australasian COVID-19 Trial (ASCOT) ADAptive Platform Trial
Acronym: ASCOT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: The Peter Doherty Institute for Infection and Immunity (Other); Australasian Society for Infectious Diseases (Other); Hunter Medical Research Institute (Unknown); Aotearoa Clinical Trials (Unknown); Australian and New Zealand Intensive Care Research Centre (Other)
Responsible Party: Principal Investigator, Associate Professor Steven Tong, Associate Professor, University of Melbourne
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: X20-0159
Record Dates: First submitted 2020-07-22; First posted 2020-07-23 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: SARS-CoV-2 Infection (COVID-19)
MeSH Terms: conditions — COVID-19 | interventions — nafamostat; Enoxaparin; Dalteparin; Tinzaparin; nirmatrelvir and ritonavir drug combination; remdesivir

STUDY DESIGN:
Intervention Model Description: Participants enrolled into the study have the option of deciding whether to be randomised in one or more (if available) treatment domains concurrently, if they meet the eligibility criteria.
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (11):
- (Arm Closed) Antiviral - Standard of care (No Intervention): Standard of care without nafamostat mesilate
- (Arm Closed) Antiviral - nafamostat mesilate (Experimental): Nafamostat continuous IV infusion for 7 days or until day of hospital discharge at a dose of 0.2mg/kg/hour. No adjustment in dose is needed for renal impairment, including for renal dialysis. The daily dose of nafamostat should be administered in 500 mL (rate of infusion 20.8 mL/hour) of normal saline. Normal saline is recommended (due to the tendency for patients with COVID-19 towards hyponatraemia) but not mandated, and 5% dextrose would be acceptable if felt clinically appropriate.
  Interventions: Drug: (Arm Closed) Nafamostat Mesilate
- (Arm Closed) Anticoagulation - standard dose thromboprophylaxis (Active Comparator): Patients will be administered a standard thromboprophylactic dose of low molecular weight heparin, choice of agent according to availability and local practice at the participating site.
  Interventions: Drug: (Arm Closed) Enoxaparin; Drug: (Arm Closed) Dalteparin; Drug: (Arm Closed) Tinzaparin
- (Arm Closed) Anticoagulation - intermediate dose thromboprophylaxis (Experimental): Patients will be administered an intermediate dose of low molecular weight heparin, choice of agent according to availability and local practice at the participating site. The maximum dose of enoxaparin will be 120 mg/d, tinzaparin 125 IU/kg/day (not available within Australia), and Dalteparin 15,000 IU/d.
  Interventions: Drug: (Arm Closed) Enoxaparin; Drug: (Arm Closed) Dalteparin; Drug: (Arm Closed) Tinzaparin
- (Arm Closed) Anticoagulation - therapeutic anticoagulation (Experimental): Therapeutic anticoagulation administered with LMWH daily until hospital discharge, admission to ICU or for a maximum of 28 days from randomisation. Choice of LMWH according to availability and local practice at the participating site
  Interventions: Drug: (Arm Closed) Enoxaparin; Drug: (Arm Closed) Dalteparin; Drug: (Arm Closed) Tinzaparin
- (Arm Never Opened) Antibody - Standard of Care (No Intervention): No hyperimmune globulin
- (Arm Never Opened) Antibody - hyperimmune globulin (Experimental): 2 doses of 30mL (3x10mL vials) of COVID-19 Hyper-Immunoglobulin (Human) given over 2 days within 48 hours of randomisation
  Interventions: Biological: (Arm Never Opened) Hyperimmune globulin
- Antiviral II - No antiviral agent (No Intervention): Participants will receive no antiviral agents intended to be active against SARS-CoV-2 for 28 days or until hospital discharge, whichever occurs first.
- Antiviral II - Nirmatrelvir-ritonavir (Experimental): The dose of nirmatrelvir-ritonavir is dependent on renal function. Participants will receive 100mg BD oral/enteral Ritonavir and either 150mg BD (if eGFR 30-59 mL/min/1.73m2) or 300mg BD (eGFR >= 60 mL/min/1.73m2) oral/enteral Nirmatrelvir. Investigators are advised to consider withholding treatment if the participant's eGFR < 30 mL/min/1.73m2.
  Interventions: Drug: Nirmatrelvir-Ritonavir
- Antiviral II - Remdisivir (Experimental): The dose of intravenous remdesivir is 200 mg on day 1 followed by 100 mg daily for a further four doses (i.e., for five doses in total) or until hospital discharge, whichever occurs first. Remdesivir will be administered as an intravenous infusion via a central or peripheral venous catheter over a 30-120 minute period, as per local practice.
  Interventions: Drug: Remdesivir
- Antiviral II - Nirmatrelvir-ritonavir + remdesivir (Experimental): Participants will receive both nirmatrelvir-ritonavir and remdesivir using the dose and administration methods described above.
  Interventions: Drug: Nirmatrelvir-Ritonavir; Drug: Remdesivir

INTERVENTIONS:
Drug: (Arm Closed) Nafamostat Mesilate — Nafamostat continuous IV infusion for 7 days or until day of hospital discharge at a dose of 0.2mg/kg/hour. No adjustment in dose is needed for renal impairment, including for renal dialysis. The daily dose of nafamostat should be administered in 500 mL (rate of infusion 20.8 mL/hour) of normal saline. Normal saline is recommended (due to the tendency for patients with COVID-19 towards hyponatraemia) but not mandated, and 5% dextrose would be acceptable if felt clinically appropriate.
  Other Names: Nafabelltan
  Arms: (Arm Closed) Antiviral - nafamostat mesilate
Drug: (Arm Closed) Enoxaparin — Patients will be administered either a standard dose, intermediate dose or therapeutic anticoagulation of low molecular weight heparin (depending on assigned arm), choice of agent according to availability and local practice at the participating site.
  The maximum dose of Enoxaparin will be 1mg/kg q12h or 1.5mg/kg q24h.
  Arms: (Arm Closed) Anticoagulation - intermediate dose thromboprophylaxis; (Arm Closed) Anticoagulation - standard dose thromboprophylaxis; (Arm Closed) Anticoagulation - therapeutic anticoagulation
Drug: (Arm Closed) Dalteparin — Patients will be administered either a standard dose, intermediate dose or therapeutic anticoagulation of low molecular weight heparin (depending on assigned arm), choice of agent according to availability and local practice at the participating site.
  The maximum dose of Dalteparin will be 100IU/kg q12h or 200IU/kg q24h.
  Arms: (Arm Closed) Anticoagulation - intermediate dose thromboprophylaxis; (Arm Closed) Anticoagulation - standard dose thromboprophylaxis; (Arm Closed) Anticoagulation - therapeutic anticoagulation
Drug: (Arm Closed) Tinzaparin — Patients will be administered either a standard dose, intermediate dose or therapeutic anticoagulation of low molecular weight heparin (depending on assigned arm), choice of agent according to availability and local practice at the participating site.
  The maximum dose of Tinzaparin will be 175IU/kg q24h (not available within Australia).
  Arms: (Arm Closed) Anticoagulation - intermediate dose thromboprophylaxis; (Arm Closed) Anticoagulation - standard dose thromboprophylaxis; (Arm Closed) Anticoagulation - therapeutic anticoagulation
Biological: (Arm Never Opened) Hyperimmune globulin — 2 doses of 30mL (3x10mL vials) of COVID-19 Hyper-Immunoglobulin (Human) given over 2 days within 48 hours of randomisation. Three vials will have approximately 10500 AU of neutralising antibodies, equivalent to approximately 200mL of convalescent plasma
  Arms: (Arm Never Opened) Antibody - hyperimmune globulin
Drug: Nirmatrelvir-Ritonavir — The dose of nirmatrelvir-ritonavir is dependent on renal function. Participants will receive 100mg BD of Ritonavir and either 150mg BD (if eGFR 30-59 mL/min/1.73m2) or 300mg BD (eGFR = 60 mL/min/1.73m2) of Nirmatrelvir. Investigators are advised to consider withholding treatment if participant's eGFR < 30 mL/min/1.73m2.
  Other Names: Paxlovid
  Arms: Antiviral II - Nirmatrelvir-ritonavir; Antiviral II - Nirmatrelvir-ritonavir + remdesivir
Drug: Remdesivir — The dose of intravenous remdesivir is 200 mg on day 1 followed by 100 mg daily for a further four doses (i.e., for five doses in total) or until hospital discharge, whichever occurs first. Remdesivir will be administered as an intravenous infusion via a central or peripheral venous catheter over a 30-120 minute period, as per local practice.
  Other Names: Veklury
  Arms: Antiviral II - Nirmatrelvir-ritonavir + remdesivir; Antiviral II - Remdisivir

SUMMARY:
An International Multi-Centre Randomised Adaptive Platform Clinical Trial to Assess the Clinical, Virological and Immunological Outcomes in Patients with SARS-CoV-2 Infection (COVID-19).

DETAILED DESCRIPTION:
ASCOT is an investigator-initiated, multi-centre, open-label, randomised controlled, Bayesian, adaptive platform trial. The objective of ASCOT is to identify the regimen (combination of interventions) associated with the highest chance of improving clinical outcomes in adults hospitalised with COVID-19.

Platform trials allow multiple questions to be evaluated simultaneously and sequentially within the platform, and evaluate interaction between different treatment options, to achieve the goal of determining the optimal combination of treatments for the disease as rapidly as possible. Study treatments are categorised into different treatment domains.

The adaptive nature of the trial means treatments within a domain or an entire domain can be removed or added based on accruing data analysed at frequent intervals or based on external evidence.

[Domain Closed] Intervention domain A (antiviral): Participants will be randomised to receive either i) standard of care without nafamostat; or ii) standard of care with nafamostat

[Never Opened] Intervention domain B (antibody): Participants will be randomised to receive either i) standard of care without hyperimmune globulin; or ii) standard of care with hyperimmune globulin

[Domain Closed] Intervention domain C (anticoagulation): Participants will be randomised to receive either i) standard dose thromboprophylaxis; or ii) intermediate dose thromboprophylaxis; or iii) therapeutic anticoagulation

Intervention domain Q (Antiviral II):

Participants will be randomised to receive either i) no antiviral agents; or ii) oral nirmatrelvir-ritonavir; or iii) intravenous remdesivir iiii) oral nirmatrelvir-ritonavir + Intravenous remdesivir

ELIGIBILITY:
Inclusion Criteria:

A.Core Platform (all participants must meet the following):

1. Adult (as defined by local jurisdiction) patient admitted to hospital with acute illness and suspected or proven SARS-CoV-2 infection.

B. Antiviral II Domain (all participants in the Antiviral II domain must meet the following):

1. SARS-CoV-2 infection has been confirmed by positive rapid antigen test OR polymerase chain reaction test within the last 7 days

Exclusion Criteria:

A. Core platform exclusions (all participants must not meet the following):

1. Death is deemed to be imminent and inevitable during the next 24 hours AND one or more of the patient, substitute decision maker or attending physician are not committed to full active treatment
2. Patient is expected to be discharged from hospital today or tomorrow
3. More than 14 days have elapsed while admitted to hospital with symptoms of an acute illness due to proven SARS-CoV-2 infection
4. Previous participation in this trial, or another trial that is analysed within the same statistical model as this trial, within the last 90 days

B. Antiviral II Domain exclusions (patients at sites participating in the Antiviral II Domain must not meet the following):

1. Severe renal impairment, defined as eGFR<30ml/min or receipt of renal replacement therapy
2. Severe hepatic impairment, defined as proven or suspected cirrhosis with Child Pugh class of C, OR acute hepatitis, defined as AST or ALT>5 times the upper limit of normal in the testing laboratory.
3. The patient has received, at the time of eligibility assessment, >24h of an antiviral agent intended to have activity against SARS-CoV-2, within the past 7 days
4. The patient is known to be pregnant or breastfeeding
5. The treating clinician believes that participation in the domain would not be in the best interests of the patient

B.1. Antiviral II Domain Non-Immune Suppressed Stratum-specific Exclusion Criteria (all non-immune suppressed patients at sites participating in the Antiviral II Domain must not meet the following):

1. Onset of COVID-related symptoms was more than 7 days (i.e., 168 hours) ago

B2. Antiviral II domain Intervention-specific Exclusion Criteria (All patients at sites participating in the Antiviral II Domain will be excluded from the below interventions if they meet the following):

Will be excluded from receiving Remdesivir if:

1. No venous access is available and none can be created
2. Known hypersensitivity to remdesivir or its excipients

Will be excluded from receiving Nirmatrelvir/ritonavir if:

1. The patient is unable to take, tolerate or absorb oral or enteral medications
2. Known hypersensitivity to any of nirmatrelvir, ritonavir or its excipients
3. Receipt of a concomitant drug with a high-risk interaction with nirmatrelvir-ritonavir which cannot be ceased or substituted.

Will be excluded from receiving no antiviral agent if:

1. The patient is in the Immune Suppressed Stratum
2. The patient is receiving or has received supplemental oxygen on the calendar day of eligibility assessment.
3. The patient is considered by the treating clinician to be at very high risk for progression to severe COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
A hierarchical ordinal scale that is a composite of mortality during the acute hospital admission and the duration of organ failure support while admitted to an ICU up until the end of study day 21. | Day 21
  * All patients who die before discharge from an acute hospital, irrespective of whether this occurs before or after day 21, will be coded as -1.
  * Survivors who receive organ failure support while admitted to an ICU within 21 days are assigned a score from 0 to 21 calculated as whole or part study days for which the patient is alive and not receiving organ failure support while admitted to an ICU up until the end of study day 21.
  * Survivors who never receive organ failure support while admitted to an ICU before the end of study day 21 will be coded as 22.

SECONDARY OUTCOMES:
Core Secondary Outcome: WHO 8-point ordinal outcome scale | Day 14
  All participants in the platform will be assessed for this outcome.
  The modified ordinal score is:
  1. Not hospitalised
  2. Hospitalised
  3. Hospitalised, requiring supplemental oxygen
  4. Hospitalised, on non-invasive ventilation or high flow oxygen devices
  5. Hospitalised, on invasive mechanical ventilation or ECMO
  6. Death
  Note. Admission to a Hospital in the Home unit is not counted as hospitalisation for the purposes of this ordinal scale. Patients who have been admitted to hospital and transferred to a Hospital in the Home unit will be assessed as either ordinal score 1 or 2.
Core Secondary Outcome: All-cause mortality | Day 28, 90 and 180
  All participants in the platform will be assessed for this outcome.
  All-cause mortality
Core Secondary Outcome: Days alive and free of hospital | Day 28
  All participants in the platform will be assessed for this outcome.
  Days alive and free of hospital, as it applies to the index hospital admission, by 28 days after randomisation
  Note 1. Days spent in a Hospital in the Home unit will not be counted as days in hospital as hospital means 'acute-care hospital' for the purposes of this endpoint.
  Note 2. If patient is discharged prior to day 28, it will be assumed the patient has not been readmitted to hospital.
Core Secondary Outcome: Days alive and free of supplemental oxygen, invasive or non-invasive ventilation | Day 28
  All participants in the platform will be assessed for this outcome.
  Number of days alive and free of supplemental oxygen, invasive or non-invasive ventilation by 28 days after randomisation
  Note. If patient is discharged prior to day 28, it will be assumed that they have not received any supplemental oxygen, invasive or non-invasive ventilation since discharge.
Core Secondary Outcome: Days alive and free of invasive or non-invasive ventilation or high flow oxygen | Day 28
  All participants in the platform will be assessed for this outcome.
  Days alive and free of invasive or non-invasive ventilation or high flow oxygen by 28 days after randomisation.
  Note. If patient is discharged prior to day 28, it will be assumed that they have not received any invasive or non-invasive ventilation since discharge
Core Secondary Outcome: Days alive and free of invasive mechanical ventilation | Day 28
  All participants in the platform will be assessed for this outcome.
  Days alive and free of invasive mechanical ventilation by 28 days after randomisation
  Note. If patient is discharged prior to day 28, it will be assumed that they have not received any invasive ventilation since discharge.
Core Secondary Outcome: Shortness of breath | Day 180
  All participants in the platform will be assessed for this outcome.
  A) Dichotomous comparison of a subjective measure of shortness of breath such as: "Are you currently experiencing shortness of breath that you didn't have before you got COVID, or which is worse now than before you got COVID?"
  B) Ordinal comparison of the modified Medical Research Council (mMRC) breathlessness scale:
  0 - I only get breathless with strenuous exercise
  1. - I get short of breath when hurrying on level ground or walking up a slight hill
  2. - On level ground, I walk slower than people of the same age because of breathlessness, or I have to stop for breath when walking at my own pace on the level
  3. - I stop for breath after walking about 100 metres or after a few minutes on level ground
  4. - I am too breathless to leave the house or I am breathless when
Core Secondary Outcome: Quality of life | Day 180
  All participants in the platform will be assessed for this outcome.
  Measured by the EQ-5D-5L questionnaire
Core Secondary Outcome: Destination at time of hospital discharge | Up to day 90
  All participants in the platform will be assessed for this outcome.
  Destination characterised as home, rehabilitation hospital, nursing home, or long-term care facility, or another acute hospital.
Core Secondary Outcome: Admission (or re-admission) to ICU | During the participant's index hospitalisation. Up to day 90.
  All participants in the platform will be assessed for this outcome.
  Admission (or re-admission) to ICU during the index hospitalisation, censored at 90 days post-randomisation
Core secondary outcome measures for participants admitted to ICU: ICU mortality | Up to day 90
  All participants in the platform who are admitted to ICU will be assessed for this outcome.
  ICU mortality, censored at 90 days post-randomisation
Core secondary outcome measures for participants admitted to ICU: ICU length of stay | Up to day 90
  All participants in the platform who are admitted to ICU will be assessed for this outcome.
  ICU length of stay, censored at 90 days post-randomisation
Core secondary outcome measures for participants admitted to ICU: Ventilator-free days | Up to day 28
  All participants in the platform who are admitted to ICU will be assessed for this outcome.
  Number of ventilator-free days, censored at 28 days post-randomisation
Core secondary outcome measures for participants admitted to ICU: Organ failure free days | Up to day 28
  All participants in the platform who are admitted to ICU will be assessed for this outcome.
  Number of organ failure free days
Antiviral II Domain Secondary Outcome: Length of hospital stay (in days) | During the participant's index hospitalisation. Censored 90 days after enrolment.
  All participants randomised to the Antiviral II domain will be assessed for this outcome
  Number of days in hospital
Antiviral II Domain Secondary Outcome: Proportion of participants with baseline respiratory symptoms in whom all acute respiratory symptoms have resolved at study day 7 | Day 7
  All participants randomised to the Antiviral II domain will be assessed for this outcome
  Proportion of participants with baseline respiratory symptoms in whom all acute respiratory symptoms have resolved at study day 7 after randomisation.
  Note 1. Respiratory symptoms are defined as one or more of: cough, sore throat, runny nose sneezing, shortness of breath or chest pain. "Acute" means the symptom in question is not usually present in that individual, or during the current COVID episode was substantially worse or more frequent than usual.
  Note 2. Resolution of all acute respiratory symptoms means return to baseline state - not necessarily the absence of all respiratory symptoms. Note 3. Ongoing non-respiratory symptoms (such as fatigue, anorexia, delirium, diarrhea) are not counted as part of this endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Tong, Prof, Study Chair — Melbourne Health
Locations (25):
- Australia (25):
  - Blacktown Hospital, Blacktown, New South Wales
  - Campbelltown Hospital, Campbelltown, New South Wales
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Wagga Wagga Base Hospital, Wagga Wagga, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Royal Darwin Hospital, Tiwi, Northern Territory
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Ballarat Health Services, Ballarat Central, Victoria
  - Eastern Health (Box Hill Hospital), Box Hill, Victoria
  - Monash Health, Clayton, Victoria
  - Northern Health, Epping, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Western Health, St Albans, Victoria
  - West Gippsland Hospital, Warragul, Victoria
  - Royal Perth Hospital, Perth, Western Australia

REFERENCES:
- [Derived] Morpeth SC, Venkatesh B, Totterdell JA, McPhee GM, Mahar RK, Jones M, Bandara M, Barina LA, Basnet BK, Bowen AC, Burke AJ, Cochrane B, Denholm JT, Dhungana A, Dore GJ, Dotel R, Duffy E, Dummer J, Foo H, Gilbey TL, Hammond NE, Hudson BJ, Jha V, Jevaji PR, John O, Joshi R, Kang G, Kaur B, Kim S, Das SK, Lau JSY, Littleford R, Marsh JA, Marschner IC, Matthews G, Maze MJ, McArthur CJ, McFadyen JD, McMahon JH, McQuilten ZK, Molton J, Mora JM, Mudaliar V, Nguyen V, O'Sullivan MVN, Pant S, Park JE, Paterson DL, Price DJ, Raymond N, Rees MA, Robinson JO, Rogers BA, Ryu WS, Sasadeusz J, Shum O, Snelling TL, Sommerville C, Trask N, Lewin SR, Hills TE, Davis JS, Roberts JA, Tong SYC. A Randomized Trial of Nafamostat for Covid-19. NEJM Evid. 2023 Nov;2(11):EVIDoa2300132. doi: 10.1056/EVIDoa2300132. Epub 2023 Oct 18. PMID 38320527
- [Derived] McQuilten ZK, Venkatesh B, Jha V, Roberts J, Morpeth SC, Totterdell JA, McPhee GM, Abraham J, Bam N, Bandara M, Bangi AK, Barina LA, Basnet BK, Bhally H, Bhusal KR, Bogati U, Bowen AC, Burke AJ, Christopher DJ, Chunilal SD, Cochrane B, Curnow JL, Das SK, Dhungana A, Di Tanna GL, Dotel R, DSouza H, Dummer J, Dutta S, Foo H, Gilbey TL, Giles ML, Goli K, Gordon A, Gyanwali P, Haksar D, Hudson BJ, Jani MK, Jevaji PR, Jhawar S, Jindal A, John MJ, John M, John FB, John O, Jones M, Joshi RD, Kamath P, Kang G, Karki AR, Karmalkar AM, Kaur B, Koganti KC, Koshy JM, Krishnamurthy MS, Lau JS, Lewin SR, Lim LL, Marschner IC, Marsh JA, Maze MJ, McGree JM, McMahon JH, Medcalf RL, Merriman EG, Misal AP, Mora JM, Mudaliar VK, Nguyen V, O'Sullivan MV, Pant S, Pant P, Paterson DL, Price DJ, Rees MA, Robinson JO, Rogers BA, Samuel S, Sasadeusz J, Sharma D, Sharma PK, Shrestha R, Shrestha SK, Shrestha P, Shukla U, Shum O, Sommerville C, Spelman T, Sullivan RP, Thatavarthi U, Tran HA, Trask N, Whitehead CL, Mahar RK, Hammond NE, McFadyen JD, Snelling TL, Davis JS, Denholm JT, Tong SYC. Anticoagulation Strategies in Non-Critically Ill Patients with Covid-19. NEJM Evid. 2023 Feb;2(2):EVIDoa2200293. doi: 10.1056/EVIDoa2200293. Epub 2022 Dec 10. PMID 38320033
- [Derived] Denholm JT, Venkatesh B, Davis J, Bowen AC, Hammond NE, Jha V, McPhee G, McQuilten Z, O'Sullivan MVN, Paterson D, Price D, Rees M, Roberts J, Jones M, Totterdell J, Snelling T, Trask N, Morpeth S, Tong SY; ASCOT ADAPT investigators. ASCOT ADAPT study of COVID-19 therapeutics in hospitalised patients: an international multicentre adaptive platform trial. Trials. 2022 Dec 14;23(1):1014. doi: 10.1186/s13063-022-06929-y. PMID 36514143
- [Derived] Bassi A, Arfin S, Joshi R, Bathla N, Hammond NE, Rajbhandari D, Tirupakuzhi Vijayaraghavan BK, Venkatesh B, Jha V. Challenges in operationalising clinical trials in India during the COVID-19 pandemic. Lancet Glob Health. 2022 Mar;10(3):e317-e319. doi: 10.1016/S2214-109X(21)00546-5. Epub 2021 Dec 22. No abstract available. PMID 34953516